CLINICAL TRIAL: NCT02355665
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group Study Using a Naturalistic Clinical Model to Measure the Efficacy and Safety of a Novel Nicotine Replacement Therapy in Smokers Motivated to Quit
Brief Title: Study to Determine the Efficacy and Safety of a Novel Nicotine Replacement Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McNeil Consumer Healthcare Division of McNEIL-PPC, Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry); McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CO-140121222102-SCCT
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine (Experimental): Nicotine Spray
  Interventions: Drug: Nicotine Spray
- Placebo (Placebo Comparator): Placebo to match Nicotine spray
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nicotine Spray — Nicotine Spray
  Arms: Nicotine
Drug: Placebo — Placebo to match nicotine spray
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of a novel nicotine product for continuous abstinence from smoking. Efficacy of product will be evaluated by assessments of self-reported abstinence, verified by exhaled carbon monoxide (CO) levels.

ELIGIBILITY:
Inclusion Criteria:

Subjects must be males or females 18-85 years of age who currently smoke cigarettes daily and are willing to stop smoking

Exclusion Criteria:

History of cardiovascular disease, stomach ulcer or diabetes unless physician's written approval is obtained.

Use of other forms of tobacco/nicotine containing products other than cigarettes within 30 days before baseline visit.

Use of nicotine replacement therapies or other smoking cessation medicines/non-drug therapies within 30 days before the baseline visit.

Pregnancy or intending to become pregnant.

Hypersensitivity to the product, history of alcohol or substance abuse.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1198 (Actual)
Dates: Start 2015-01-31 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2016-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Myers, MD, Study Director — McNeil Consumer Healthcare Division of McNEIL-PPC, Inc.
Locations (8):
- United States (8):
  - Mayo Clinic, Scottsdale, Arizona
  - Los Angeles Clinical Trials, Burbank, California
  - Radiant Research, Inc, Chicago, Illinois
  - University of Maryland, College Park, Maryland
  - Radiant Research, Inc., Akron, Ohio
  - Radiant Research, Cincinnati, Ohio
  - Radiant Research, Inc, Dallas, Texas
  - Radiant Research, Inc, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nides M, Danielsson T, Saunders F, Perfekt R, Kapikian R, Solla J, Leischow SJ, Myers A. Efficacy and Safety of a Nicotine Mouth Spray for Smoking Cessation: A Randomized, Multicenter, Controlled Study in a Naturalistic Setting. Nicotine Tob Res. 2020 Mar 16;22(3):339-345. doi: 10.1093/ntr/nty246. PMID 30452732

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo capsaicin mouth spray, 0 mg nicotine/dose, intraorally per label directions
- Nicotine: Nicotine mouth spray, 1 mg nicotine/dose, intraorally per label directions
Period: Overall Study
Arm/Group | Placebo | Nicotine
Started | 601 | 597
Completed | 352 | 365
Not Completed | 249 | 232
Not completed — Adverse Event | 16 | 24
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 90 | 100
Not completed — Lost to Follow-up | 131 | 103
Not completed — Death | 4 | 2
Not completed — Compliance, PI decision, move, eligible | 6 | 3

BASELINE CHARACTERISTICS:
Population: Analysis was based on the Full Analysis Set which included all study participants randomly assigned to study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nicotine | Total
Number analyzed (Participants) | 601 | 597 | 1198
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (11.72) | 51.5 (11.7) | 51.3 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 319 | 332 | 651
  Male | 282 | 265 | 547
Region of Enrollment [Count of Participants; unit: Participants]
  United States: USA | 601 | 597 | 1198

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Continuous Smoking Abstinence From Week 2 to Week 6
Description: Percentage of participants with carbon monoxide (CO)-verified self-report of continuous abstinence from smoking
Time Frame: Week 2 to Week 6
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 601 | 597
Percentage of Participants | 2.5 | 5.0
Statistical Analysis 1: Comparison: Placebo vs Nicotine; The null hypothesis was no difference in continuous smoking abstinence rates between treatments. The alternative hypothesis was a difference in continuous smoking abstinence rates between treatments; Test type: Superiority; p = 0.021, Cochran-Mantel-Haenszel — The significance threshold level was 0.05 (two-sided); Cochran-Mantel-Haenszel test stratified by study site and number of cigarettes smoked per day at baseline (<20 per day vs ≥20 per day); Estimated Success Rate Ratio = 2.00, 95% CI 2-sided [1.10 to 3.66] — Estimated Success Rate Ratio = Nicotine/Placebo

2. Secondary Outcome: Percentage of Participants With Continuous Smoking Abstinence From Week 2 to Week 12
Description: Percentage of participants with carbon monoxide (CO)-verified self-report of continuous abstinence from smoking
Time Frame: Week 2 to Week 12
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 601 | 597
Percentage of Participants | 1.3 | 4.0
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 1, analysis 1]; Estimated Success Rate Ratio = 3.04, 95% CI 2-sided [1.39 to 6.68] — Estimated Success Rate Ratio = Nicotine/Placebo

3. Secondary Outcome: Percentage of Participants With Continuous Smoking Abstinence From Week 2 to Week 26
Description: Percentage of participants with carbon monoxide (CO)-verified self-report of continuous abstinence from smoking
Time Frame: Week 2 to Week 26
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 601 | 597
Percentage of Participants | 1.2 | 3.4
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.011, Cochran-Mantel-Haenszel — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 1, analysis 1]; Estimated Success Rate Ratio = 2.87, 95% CI 2-sided [1.23 to 6.71] — Estimated Success Rate Ratio = Nicotine/Placebo

4. Secondary Outcome: Percentage of Participants With Continuous Smoking Abstinence From Week 2 to Week 4
Description: Percentage of participants with carbon monoxide (CO)-verified self-report of continuous abstinence from smoking
Time Frame: Week 2 to Week 4
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 601 | 597
Percentage of Participants | 4.0 | 6.7
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.040, Cochran-Mantel-Haenszel — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 1, analysis 1]; Estimated Success Rate Ratio = 1.66, 95% CI 2-sided [1.02 to 2.71] — Estimated Success Rate Ratio = Nicotine/Placebo

5. Secondary Outcome: Percentage of Participants With Continuous Smoking Abstinence From Week 2 to Week 8
Description: Percentage of participants with carbon monoxide (CO)-verified self-report of continuous abstinence from smoking
Time Frame: Week 2 to Week 8
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 601 | 597
Percentage of Participants | 2.2 | 4.5
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.023, Cochran-Mantel-Haenszel — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 1, analysis 1]; Estimated Success Rate Ratio = 2.09, 95% CI 2-sided [1.09 to 3.98] — Estimated Success Rate Ratio = Nicotine/Placebo

6. Secondary Outcome: Percentage of Participants With Continuous Smoking Abstinence From Week 2 to Week 16
Description: Percentage of participants with carbon monoxide (CO)-verified self-report of continuous abstinence from smoking
Time Frame: Week 2 to Week 16
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 601 | 597
Percentage of Participants | 1.3 | 3.9
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 1, analysis 1]; Estimated Success Rate Ratio = 2.91, 95% CI 2-sided [1.32 to 6.42] — Estimated Success Rate Ratio = Nicotine/Placebo

7. Secondary Outcome: Percentage of Participants With Continuous Smoking Abstinence From Week 2 to Week 20
Description: Percentage of participants with carbon monoxide (CO)-verified self-report of continuous abstinence from smoking
Time Frame: Week 2 to Week 20
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 601 | 597
Percentage of Participants | 1.3 | 3.5
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.013, Cochran-Mantel-Haenszel — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 1, analysis 1]; Estimated Success Rate Ratio = 2.66, 95% CI 2-sided [1.20 to 5.92] — Estimated Success Rate Ratio = Nicotine/Placebo

8. Secondary Outcome: Percentage Distribution of the Rating of Desire/Urge to Smoke on a Categorical Scale at Week 1
Description: Participants were asked if during the last 24 hours they experienced the desire/urge to smoke on a 5-grade categorical scale of 0 - 4 (where 0=not at all and 4=extremely so).
Time Frame: Week 1
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 21 | 39
Percentage of Participants
  Not at all (0) | 9.5 | 12.8
  Somewhat (1) | 33.3 | 35.9
  Moderately so (2) | 33.3 | 25.6
  Very much so (3) | 19.0 | 15.4
  Extremely so (4) | 4.8 | 10.3
Statistical Analysis 1: Comparison: Placebo vs Nicotine; The null hypothesis was no difference in distribution of the ratings of desire/urge to smoke between treatments. The alternative hypothesis was a difference in distribution of the ratings of desire/urge to smoke between treatments; Test type: Superiority; p = 0.847, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.02, 95% CI 2-sided [-0.64 to 0.60] — Estimated Mean Difference = Nicotine - Placebo

9. Secondary Outcome: Percentage Distribution of the Rating of Desire/Urge to Smoke on a Categorical Scale at Week 2
Description: as for outcome 8
Time Frame: Week 2
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 25 | 58
Percentage of Participants
  Not at all (0) | 24.0 | 15.5
  Somewhat (1) | 28.0 | 36.2
  Moderately so (2) | 20.0 | 34.5
  Very much so (3) | 20.0 | 10.3
  Extremely so (4) | 8.0 | 3.4
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.861, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.10, 95% CI 2-sided [-0.62 to 0.42] — Estimated Mean Difference = Nicotine - Placebo

10. Secondary Outcome: Percentage Distribution of the Rating of Desire/Urge to Smoke on a Categorical Scale at Week 4
Description: as for outcome 8
Time Frame: Week 4
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 26 | 43
Percentage of Participants
  Not at all (0) | 19.2 | 37.2
  Somewhat (1) | 53.8 | 39.5
  Moderately so (2) | 23.1 | 16.3
  Very much so (3) | 3.8 | 7.0
  Extremely so (4) | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.266, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.19, 95% CI 2-sided [-0.61 to 0.24] — Estimated Mean Difference = Nicotine - Placebo

11. Secondary Outcome: Percentage Distribution of the Rating of Desire/Urge to Smoke on a Categorical Scale at Week 6
Description: as for outcome 8
Time Frame: Week 6
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 32 | 54
Percentage of Participants
  Not at all (0) | 43.8 | 31.5
  Somewhat (1) | 31.3 | 42.6
  Moderately so (2) | 12.5 | 18.5
  Very much so (3) | 9.4 | 3.7
  Extremely so (4) | 3.1 | 3.7
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.487, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = 0.09, 95% CI 2-sided [-0.38 to 0.55] — Estimated Mean Difference = Nicotine - Placebo

12. Secondary Outcome: Percentage Distribution of the Rating of Irritability/Frustration/Anger on a Categorical Scale at Week 1
Description: Participants were asked if during the last 24 hours they experienced irritability/frustration/anger on a 5-grade categorical scale of 0 - 4 (where 0=not at all and 4=extremely so).
Time Frame: Week 1
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 21 | 39
Percentage of Participants
  Not at all (0) | 38.1 | 51.3
  Somewhat (1) | 38.1 | 28.2
  Moderately so (2) | 19.0 | 15.4
  Very much so (3) | 4.8 | 0.0
  Extremely so (4) | 0.0 | 5.1
Statistical Analysis 1: Comparison: Placebo vs Nicotine; The null hypothesis was no difference in distribution of the ratings of irritability/frustration/anger between treatments. The alternative hypothesis was a difference in distribution of the ratings of irritability/frustration/anger between treatments; Test type: Superiority; p = 0.433, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.11, 95% CI 2-sided [-0.65 to 0.43] — Estimated Mean Difference = Nicotine - Placebo

13. Secondary Outcome: Percentage Distribution of the Rating of Irritability/Frustration/Anger on a Categorical Scale at Week 2
Description: as for outcome 12
Time Frame: Week 2
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 25 | 58
Percentage of Participants
  Not at all (0) | 28.0 | 56.9
  Somewhat (1) | 40.0 | 24.1
  Moderately so (2) | 12.0 | 8.6
  Very much so (3) | 8.0 | 5.2
  Extremely so (4) | 12.0 | 5.2
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.022, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.58, 95% CI 2-sided [-1.15 to -0.01] — Estimated Mean Difference = Nicotine - Placebo

14. Secondary Outcome: Percentage Distribution of the Rating of Irritability/Frustration/Anger on a Categorical Scale at Week 4
Description: as for outcome 12
Time Frame: Week 4
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 26 | 43
Percentage of Participants
  Not at all (0) | 46.2 | 55.8
  Somewhat (1) | 34.6 | 23.3
  Moderately so (2) | 15.4 | 11.6
  Very much so (3) | 3.8 | 7.0
  Extremely so (4) | 0.0 | 2.3
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.665, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.00, 95% CI 2-sided [-0.50 to 0.49] — Estimated Mean Difference = Nicotine - Placebo

15. Secondary Outcome: Percentage Distribution of the Rating of Irritability/Frustration/Anger on a Categorical Scale at Week 6
Description: as for outcome 12
Time Frame: Week 6
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 32 | 54
Percentage of Participants
  Not at all (0) | 43.8 | 61.1
  Somewhat (1) | 43.8 | 20.4
  Moderately so (2) | 6.3 | 13.0
  Very much so (3) | 6.3 | 3.7
  Extremely so (4) | 0.0 | 1.9
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.300, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.10, 95% CI 2-sided [-0.51 to 0.31] — Estimated Mean Difference = Nicotine - Placebo

16. Secondary Outcome: Percentage Distribution of the Rating of Restlessness on a Categorical Scale at Week 1
Description: Participants were asked if during the last 24 hours they experienced restlessness on a 5-grade categorical scale of 0 - 4 (where 0=not at all and 4=extremely so).
Time Frame: Week 1
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 21 | 39
Percentage of Participants
  Not at all (0) | 47.6 | 43.6
  Somewhat (1) | 14.3 | 30.8
  Moderately so (2) | 23.8 | 17.9
  Very much so (3) | 9.5 | 5.1
  Extremely so (4) | 4.8 | 2.6
Statistical Analysis 1: Comparison: Placebo vs Nicotine; The null hypothesis was no difference in distribution of the ratings of restlessness between treatments. The alternative hypothesis was a difference in distribution of the ratings of restlessness between treatments; Test type: Superiority; p = 0.754, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.17, 95% CI 2-sided [-0.78 to 0.43] — Estimated Mean Difference = Nicotine - Placebo

17. Secondary Outcome: Percentage Distribution of the Rating of Restlessness on a Categorical Scale at Week 2
Description: as for outcome 16
Time Frame: Week 2
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 25 | 58
Percentage of Participants
  Not at all (0) | 40.0 | 58.6
  Somewhat (1) | 32.0 | 20.7
  Moderately so (2) | 12.0 | 17.2
  Very much so (3) | 12.0 | 1.7
  Extremely so (4) | 4.0 | 1.7
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.116, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.41, 95% CI 2-sided [-0.89 to 0.08] — Estimated Mean Difference = Nicotine - Placebo

18. Secondary Outcome: Percentage Distribution of the Rating of Restlessness on a Categorical Scale at Week 4
Description: as for outcome 16
Time Frame: Week 4
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 26 | 43
Percentage of Participants
  Not at all (0) | 53.8 | 62.8
  Somewhat (1) | 34.6 | 32.6
  Moderately so (2) | 11.5 | 2.3
  Very much so (3) | 0.0 | 2.3
  Extremely so (4) | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.392, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.14, 95% CI 2-sided [-0.47 to 0.20] — Estimated Mean Difference = Nicotine - Placebo

19. Secondary Outcome: Percentage Distribution of the Rating of Restlessness on a Categorical Scale at Week 6
Description: as for outcome 16
Time Frame: Week 6
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 32 | 54
Percentage of Participants
  Not at all (0) | 46.9 | 63.0
  Somewhat (1) | 37.5 | 24.1
  Moderately so (2) | 9.4 | 11.1
  Very much so (3) | 6.3 | 1.9
  Extremely so (4) | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.179, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.23, 95% CI 2-sided [-0.59 to 0.13] — Estimated Mean Difference = Nicotine - Placebo

20. Secondary Outcome: Percentage Distribution of the Rating of Difficulty Concentrating on a Categorical Scale at Week 1
Description: Participants were asked if during the last 24 hours they experienced difficulty concentrating on a 5-grade categorical scale of 0 - 4 (where 0=not at all and 4=extremely so).
Time Frame: Week 1
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 21 | 39
Percentage of Participants
  Not at all (0) | 66.7 | 69.2
  Somewhat (1) | 23.8 | 17.9
  Moderately so (2) | 4.8 | 7.7
  Very much so (3) | 4.8 | 5.1
  Extremely so (4) | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Nicotine; The null hypothesis was no difference in distribution of the ratings of difficulty concentrating between treatments. The alternative hypothesis was a difference in distribution of the ratings of difficulty concentrating between treatments; Test type: Superiority; p = 0.925, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = 0.01, 95% CI 2-sided [-0.44 to 0.47] — Estimated Mean Difference = Nicotine - Placebo

21. Secondary Outcome: Percentage Distribution of the Rating of Difficulty Concentrating on a Categorical Scale at Week 2
Description: as for outcome 20
Time Frame: Week 2
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 25 | 58
Percentage of Participants
  Not at all (0) | 52.0 | 63.8
  Somewhat (1) | 32.0 | 24.1
  Moderately so (2) | 8.0 | 6.9
  Very much so (3) | 4.0 | 3.4
  Extremely so (4) | 4.0 | 1.7
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.325, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.21, 95% CI 2-sided [-0.66 to 0.24] — Estimated Mean Difference = Nicotine - Placebo

22. Secondary Outcome: Percentage Distribution of the Rating of Difficulty Concentrating on a Categorical Scale at Week 4
Description: as for outcome 20
Time Frame: Week 4
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 26 | 43
Percentage of Participants
  Not at all (0) | 73.1 | 74.4
  Somewhat (1) | 23.1 | 11.6
  Moderately so (2) | 3.8 | 9.3
  Very much so (3) | 0.0 | 4.7
  Extremely so (4) | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.891, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = 0.13, 95% CI 2-sided [-0.24 to 0.51] — Estimated Mean Difference = Nicotine - Placebo

23. Secondary Outcome: Percentage Distribution of the Rating of Difficulty Concentrating on a Categorical Scale at Week 6
Description: as for outcome 20
Time Frame: Week 6
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 32 | 54
Percentage of Participants
  Not at all (0) | 71.9 | 74.1
  Somewhat (1) | 12.5 | 16.7
  Moderately so (2) | 9.4 | 5.6
  Very much so (3) | 6.3 | 3.7
  Extremely so (4) | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.721, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.11, 95% CI 2-sided [-0.48 to 0.25] — Estimated Mean Difference = Nicotine - Placebo

24. Secondary Outcome: Percentage Distribution of the Rating of Anxiety on a Categorical Scale at Week 1
Description: Participants were asked if during the last 24 hours they experienced anxiety on a 5-grade categorical scale of 0 - 4 (where 0=not at all and 4=extremely so).
Time Frame: Week 1
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 21 | 39
Percentage of Participants
  Not at all (0) | 52.4 | 59.0
  Somewhat (1) | 28.6 | 28.2
  Moderately so (2) | 19.0 | 7.7
  Very much so (3) | 0.0 | 0.0
  Extremely so (4) | 0.0 | 5.1
Statistical Analysis 1: Comparison: Placebo vs Nicotine; The null hypothesis was no difference in distribution of the ratings of anxiety between treatments. The alternative hypothesis was a difference in distribution of the ratings of anxiety between treatments; Test type: Superiority; p = 0.608, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.03, 95% CI 2-sided [-0.54 to 0.49] — Estimated Mean Difference = Nicotine - Placebo

25. Secondary Outcome: Percentage Distribution of the Rating of Anxiety on a Categorical Scale at Week 2
Description: as for outcome 24
Time Frame: Week 2
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 25 | 58
Percentage of Participants
  Not at all (0) | 44.0 | 72.4
  Somewhat (1) | 24.0 | 12.1
  Moderately so (2) | 12.0 | 8.6
  Very much so (3) | 12.0 | 3.4
  Extremely so (4) | 8.0 | 3.4
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p = 0.014, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.63, 95% CI 2-sided [-1.16 to -0.09] — Estimated Mean Difference = Nicotine - Placebo

26. Secondary Outcome: Percentage Distribution of the Rating of Anxiety on a Categorical Scale at Week 4
Description: as for outcome 24
Time Frame: Week 4
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 26 | 43
Percentage of Participants
  Not at all (0) | 65.4 | 65.1
  Somewhat (1) | 26.9 | 23.3
  Moderately so (2) | 7.7 | 11.6
  Very much so (3) | 0.0 | 0.0
  Extremely so (4) | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p = 0.900, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = 0.04, 95% CI 2-sided [-0.30 to 0.38] — Estimated Mean Difference = Nicotine - Placebo

27. Secondary Outcome: Percentage Distribution of the Rating of Anxiety on a Categorical Scale at Week 6
Description: as for outcome 24
Time Frame: Week 6
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 32 | 54
Percentage of Participants
  Not at all (0) | 62.5 | 66.7
  Somewhat (1) | 25.0 | 20.4
  Moderately so (2) | 6.3 | 9.3
  Very much so (3) | 6.3 | 3.7
  Extremely so (4) | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p = 0.731, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.06, 95% CI 2-sided [-0.44 to 0.31] — Estimated Mean Difference = Nicotine - Placebo

28. Secondary Outcome: Percentage Distribution of the Rating of Dysphoric or Depressed Mood on a Categorical Scale at Week 1
Description: Participants were asked if during the last 24 hours they experienced dysphoric or depressed mood on a 5-grade categorical scale of 0 - 4 (where 0=not at all and 4=extremely so).
Time Frame: Week 1
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 21 | 39
Percentage of Participants
  Not at all (0) | 81.0 | 87.2
  Somewhat (1) | 19.0 | 5.1
  Moderately so (2) | 0.0 | 5.1
  Very much so (3) | 0.0 | 2.6
  Extremely so (4) | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Nicotine; The null hypothesis was no difference in distribution of the ratings of dysphoric or depressed mood between treatments. The alternative hypothesis was a difference in distribution of the ratings of dysphoric or depressed mood between treatments; Test type: Superiority; p = 0.635, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = 0.04, 95% CI 2-sided [-0.28 to 0.36] — Estimated Mean Difference = Nicotine - Placebo

29. Secondary Outcome: Percentage Distribution of the Rating of Dysphoric or Depressed Mood on a Categorical Scale at Week 2
Description: as for outcome 28
Time Frame: Week 2
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 25 | 58
Percentage of Participants
  Not at all (0) | 72.0 | 84.5
  Somewhat (1) | 20.0 | 5.2
  Moderately so (2) | 8.0 | 6.9
  Very much so (3) | 0.0 | 1.7
  Extremely so (4) | 0.0 | 1.7
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p = 0.273, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.05, 95% CI 2-sided [-0.42 to 0.32] — Estimated Mean Difference = Nicotine - Placebo

30. Secondary Outcome: Percentage Distribution of the Rating of Dysphoric or Depressed Mood on a Categorical Scale at Week 4
Description: as for outcome 28
Time Frame: Week 4
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 26 | 43
Percentage of Participants
  Not at all (0) | 84.6 | 86.0
  Somewhat (1) | 11.5 | 9.3
  Moderately so (2) | 0.0 | 2.3
  Very much so (3) | 0.0 | 2.3
  Extremely so (4) | 3.8 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p = 0.879, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.06, 95% CI 2-sided [-0.40 to 0.28] — Estimated Mean Difference = Nicotine - Placebo

31. Secondary Outcome: Percentage Distribution of the Rating of Dysphoric or Depressed Mood on a Categorical Scale at Week 6
Description: as for outcome 28
Time Frame: Week 6
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 32 | 54
Percentage of Participants
  Not at all (0) | 78.1 | 75.9
  Somewhat (1) | 15.6 | 16.7
  Moderately so (2) | 3.1 | 5.6
  Very much so (3) | 3.1 | 1.9
  Extremely so (4) | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p = 0.823, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = 0.02, 95% CI 2-sided [-0.28 to 0.32] — Estimated Mean Difference = Nicotine - Placebo

32. Secondary Outcome: Percentage Distribution of the Rating of Insomnia on a Categorical Scale at Week 1
Description: Participants were asked if during the last 24 hours they experienced insomnia on a 5-grade categorical scale of 0 - 4 (where 0=not at all and 4=extremely so).
Time Frame: Week 1
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 21 | 39
Percentage of Participants
  Not at all (0) | 76.2 | 79.5
  Somewhat (1) | 14.3 | 12.8
  Moderately so (2) | 9.5 | 2.6
  Very much so (3) | 0.0 | 5.1
  Extremely so (4) | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Nicotine; The null hypothesis was no difference in distribution of the ratings of insomnia between treatments. The alternative hypothesis was a difference in distribution of the ratings of insomnia between treatments; Test type: Superiority; p = 0.804, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = 0.00, 95% CI 2-sided [-0.40 to 0.40] — Estimated Mean Difference = Nicotine - Placebo

33. Secondary Outcome: Percentage Distribution of the Rating of Insomnia on a Categorical Scale at Week 2
Description: as for outcome 32
Time Frame: Week 2
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 25 | 58
Percentage of Participants
  Not at all (0) | 76.0 | 67.2
  Somewhat (1) | 16.0 | 20.7
  Moderately so (2) | 0.0 | 5.2
  Very much so (3) | 8.0 | 5.2
  Extremely so (4) | 0.0 | 1.7
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 32, analysis 1]; Test type: Superiority; p = 0.438, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = 0.13, 95% CI 2-sided [-0.30 to 0.57] — Estimated Mean Difference = Nicotine - Placebo

34. Secondary Outcome: Percentage Distribution of the Rating of Insomnia on a Categorical Scale at Week 4
Description: as for outcome 32
Time Frame: Week 4
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 26 | 43
Percentage of Participants
  Not at all (0) | 61.5 | 69.8
  Somewhat (1) | 26.9 | 20.9
  Moderately so (2) | 11.5 | 7.0
  Very much so (3) | 0.0 | 2.3
  Extremely so (4) | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 32, analysis 1]; Test type: Superiority; p = 0.517, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.08, 95% CI 2-sided [-0.44 to 0.28] — Estimated Mean Difference = Nicotine - Placebo

35. Secondary Outcome: Percentage Distribution of the Rating of Insomnia on a Categorical Scale at Week 6
Description: as for outcome 32
Time Frame: Week 6
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 32 | 54
Percentage of Participants
  Not at all (0) | 62.5 | 83.3
  Somewhat (1) | 21.9 | 11.1
  Moderately so (2) | 6.3 | 3.7
  Very much so (3) | 6.3 | 1.9
  Extremely so (4) | 3.1 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 32, analysis 1]; Test type: Superiority; p = 0.027, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.42, 95% CI 2-sided [-0.77 to -0.06] — Estimated Mean Difference = Nicotine - Placebo

36. Secondary Outcome: Percentage Distribution of the Rating of Increased Appetite on a Categorical Scale at Week 1
Description: Participants were asked if during the last 24 hours they experienced increased appetite on a 5-grade categorical scale of 0 - 4 (where 0=not at all and 4=extremely so).
Time Frame: Week 1
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 21 | 39
Percentage of Participants
  Not at all (0) | 9.5 | 43.6
  Somewhat (1) | 52.4 | 28.2
  Moderately so (2) | 23.8 | 5.1
  Very much so (3) | 14.3 | 17.9
  Extremely so (4) | 0.0 | 5.1
Statistical Analysis 1: Comparison: Placebo vs Nicotine; The null hypothesis was no difference in distribution of the ratings of increased appetite between treatments. The alternative hypothesis was a difference in distribution of the ratings of increased appetite between treatments; Test type: Superiority; p = 0.105, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.30, 95% CI 2-sided [-0.93 to 0.33] — Estimated Mean Difference = Nicotine - Placebo

37. Secondary Outcome: Percentage Distribution of the Rating of Increased Appetite on a Categorical Scale at Week 2
Description: as for outcome 36
Time Frame: Week 2
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 25 | 58
Percentage of Participants
  Not at all (0) | 28.0 | 41.4
  Somewhat (1) | 36.0 | 25.9
  Moderately so (2) | 24.0 | 12.1
  Very much so (3) | 12.0 | 17.2
  Extremely so (4) | 0.0 | 3.4
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 36, analysis 1]; Test type: Superiority; p = 0.604, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.04, 95% CI 2-sided [-0.60 to 0.51] — Estimated Mean Difference = Nicotine - Placebo

38. Secondary Outcome: Percentage Distribution of the Rating of Increased Appetite on a Categorical Scale at Week 4
Description: as for outcome 36
Time Frame: Week 4
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 26 | 43
Percentage of Participants
  Not at all (0) | 30.8 | 44.2
  Somewhat (1) | 26.9 | 30.2
  Moderately so (2) | 23.1 | 11.6
  Very much so (3) | 15.4 | 9.3
  Extremely so (4) | 3.8 | 4.7
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 36, analysis 1]; Test type: Superiority; p = 0.194, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.35, 95% CI 2-sided [-0.93 to 0.24] — Estimated Mean Difference = Nicotine - Placebo

39. Secondary Outcome: Percentage Distribution of the Rating of Increased Appetite on a Categorical Scale at Week 6
Description: as for outcome 36
Time Frame: Week 6
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 32 | 54
Percentage of Participants
  Not at all (0) | 21.9 | 35.2
  Somewhat (1) | 43.8 | 31.5
  Moderately so (2) | 18.8 | 14.8
  Very much so (3) | 12.5 | 14.8
  Extremely so (4) | 3.1 | 3.7
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 36, analysis 1]; Test type: Superiority; p = 0.502, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.11, 95% CI 2-sided [-0.62 to 0.40] — Estimated Mean Difference = Nicotine - Placebo

40. Secondary Outcome: Aggregated Withdrawal Score at Week 1
Description: Participants were asked if during the last 24 hours they experienced each of 7 withdrawal symptoms on a 5-grade categorical scale of 0 - 4 (where 0=not at all and 4=extremely so). The aggregated withdrawal symptom score was the sum of the scores of the 7 withdrawal symptoms (irritability-frustration-anger, restlessness, difficulty concentrating, anxiety, dysphoric or depressed mood, insomnia, and increased appetite). The total scores are reported with a minimum possible score of 0 and a maximum possible score of 28.
Time Frame: Week 1
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 21 | 39
units on a scale | 5.1 (4.25) | 4.5 (4.20)
Statistical Analysis 1: Comparison: Placebo vs Nicotine; The null hypothesis was no difference in distribution of aggregated withdrawal scores between treatments. The alternative hypothesis was a difference in distribution of aggregated withdrawal scores between treatments; Test type: Superiority; p = 0.483, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.56, 95% CI 2-sided [-2.84 to 1.73] — Estimated Mean Difference = Nicotine - Placebo

41. Secondary Outcome: Aggregated Withdrawal Score at Week 2
Description: as for outcome 40
Time Frame: Week 2
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 25 | 58
units on a scale | 6.3 (5.46) | 4.5 (5.02)
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 40, analysis 1]; Test type: Superiority; p = 0.102, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -1.79, 95% CI 2-sided [-4.24 to 0.67] — Estimated Mean Difference = Nicotine - Placebo

42. Secondary Outcome: Aggregated Withdrawal Score at Week 4
Description: as for outcome 40
Time Frame: Week 4
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 26 | 43
units on a scale | 4.2 (3.53) | 3.7 (3.77)
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 40, analysis 1]; Test type: Superiority; p = 0.532, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -0.45, 95% CI 2-sided [-2.27 to 1.38] — Estimated Mean Difference = Nicotine - Placebo

43. Secondary Outcome: Aggregated Withdrawal Score at Week 6
Description: as for outcome 40
Time Frame: Week 6
Population: Analysis was based on randomized participants verified abstinent from smoking since the last visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 32 | 54
units on a scale | 4.8 (5.11) | 3.8 (3.80)
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 40, analysis 1]; Test type: Superiority; p = 0.354, Wilcoxon (Mann-Whitney) — The significance threshold level was 0.05 (two-sided); Estimated Mean Difference = -1.01, 95% CI 2-sided [-2.93 to 0.91] — Estimated Mean Difference = Nicotine - Placebo

44. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 1
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 1
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 512 | 502
Number of sprays | 15.6 (10.77) | 12.3 (8.78)

45. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 2
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 2
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 492 | 486
Number of sprays | 15.7 (12.08) | 11.8 (9.19)

46. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 3
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 3
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 467 | 462
Number of sprays | 14.6 (11.15) | 11.6 (9.31)

47. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 4
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 4
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 449 | 444
Number of sprays | 13.8 (11.05) | 11.3 (10.66)

48. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 5
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 5
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 423 | 428
Number of sprays | 14.2 (12.17) | 10.9 (9.91)

49. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 6
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 6
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 406 | 412
Number of sprays | 13.1 (10.49) | 10.5 (9.71)

50. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 7
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 7
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 392 | 387
Number of sprays | 12.3 (9.63) | 9.9 (8.80)

51. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 8
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 8
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 378 | 377
Number of sprays | 12.1 (10.15) | 10.1 (8.90)

52. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 9
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 9
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 356 | 362
Number of sprays | 11.8 (9.98) | 9.7 (8.92)

53. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 10
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 10
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 336 | 337
Number of sprays | 11.6 (9.86) | 9.3 (8.66)

54. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 11
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 11
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 317 | 329
Number of sprays | 11.3 (9.80) | 8.8 (8.55)

55. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 12
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 12
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 306 | 332
Number of sprays | 9.7 (7.69) | 7.9 (7.90)

56. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 13
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 13
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 240 | 251
Number of sprays | 10.2 (8.28) | 8.4 (8.36)

57. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 14
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 14
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 223 | 237
Number of sprays | 10.3 (9.20) | 9.2 (12.88)

58. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 15
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 15
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 213 | 228
Number of sprays | 10.5 (9.66) | 8.2 (8.47)

59. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 16
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 16
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 206 | 218
Number of sprays | 9.2 (8.70) | 8.0 (8.47)

60. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 17
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 17
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 189 | 194
Number of sprays | 9.2 (8.58) | 8.0 (7.56)

61. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 18
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 18
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 182 | 192
Number of sprays | 9.4 (8.84) | 8.2 (8.80)

62. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 19
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 19
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 171 | 180
Number of sprays | 9.1 (8.49) | 8.3 (8.59)

63. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 20
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 20
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 173 | 174
Number of sprays | 7.8 (6.94) | 8.2 (8.50)

64. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 21
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 21
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 164 | 161
Number of sprays | 7.8 (7.32) | 8.2 (8.84)

65. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 22
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 22
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 155 | 158
Number of sprays | 7.5 (7.27) | 7.8 (8.32)

66. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 23
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 23
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 147 | 155
Number of sprays | 7.7 (6.97) | 7.4 (8.04)

67. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 24
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 24
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 139 | 143
Number of sprays | 7.2 (6.50) | 7.2 (8.09)

68. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 25
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 25
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 142 | 143
Number of sprays | 6.6 (6.08) | 6.7 (7.95)

69. Secondary Outcome: Total Daily Number of Self-Reported Spray Doses at Week 26
Description: Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 26
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 129 | 137
Number of sprays | 6.3 (5.91) | 6.3 (6.81)

70. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 1
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 1
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 512 | 502
Number of sprays | 22.1 (17.66) | 17.2 (11.63)

71. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 2
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 2
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 492 | 486
Number of sprays | 21.2 (16.83) | 15.4 (10.96)

72. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 3
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 3
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 467 | 462
Number of sprays | 19.2 (14.78) | 15.2 (13.51)

73. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 4
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 4
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 449 | 444
Number of sprays | 17.9 (13.58) | 15.8 (23.44)

74. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 5
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 5
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 423 | 428
Number of sprays | 19.2 (30.71) | 15.1 (27.65)

75. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 6
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 6
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 406 | 412
Number of sprays | 17.5 (14.59) | 14.6 (24.02)

76. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 7
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 7
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 392 | 387
Number of sprays | 16.0 (12.39) | 12.8 (11.57)

77. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 8
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 8
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 378 | 377
Number of sprays | 16.0 (13.05) | 13.6 (14.59)

78. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 9
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 9
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 356 | 362
Number of sprays | 15.4 (13.53) | 12.2 (11.01)

79. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 10
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 10
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 336 | 337
Number of sprays | 14.7 (12.47) | 11.4 (10.08)

80. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 11
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 11
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 317 | 329
Number of sprays | 15.1 (26.23) | 11.2 (11.35)

81. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 12
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 12
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 306 | 332
Number of sprays | 12.6 (9.70) | 9.8 (8.82)

82. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 13
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 13
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 240 | 251
Number of sprays | 12.9 (9.78) | 10.5 (9.29)

83. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 14
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 14
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 223 | 237
Number of sprays | 13.1 (10.95) | 13.6 (40.98)

84. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 15
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 15
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 213 | 228
Number of sprays | 15.3 (30.31) | 10.8 (12.53)

85. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 16
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 16
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 206 | 218
Number of sprays | 12.4 (12.80) | 10.0 (9.87)

86. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 17
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 17
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 189 | 194
Number of sprays | 11.5 (10.19) | 10.5 (9.76)

87. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 18
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 18
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 182 | 192
Number of sprays | 12.3 (11.94) | 10.3 (10.01)

88. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 19
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 19
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 171 | 180
Number of sprays | 11.2 (9.85) | 10.3 (10.20)

89. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 20
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 20
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 173 | 174
Number of sprays | 10.5 (9.38) | 10.5 (11.69)

90. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 21
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 21
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 164 | 161
Number of sprays | 10.0 (8.82) | 11.0 (13.56)

91. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 22
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 22
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 155 | 158
Number of sprays | 9.4 (8.89) | 10.8 (16.62)

92. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 23
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 23
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 147 | 155
Number of sprays | 10.5 (12.79) | 9.1 (9.33)

93. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 24
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 24
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 139 | 143
Number of sprays | 9.2 (8.50) | 8.8 (9.20)

94. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 25
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 25
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 142 | 143
Number of sprays | 8.5 (7.24) | 8.4 (9.95)

95. Secondary Outcome: Maximum Total Daily Number of Self-Reported Spray Doses at Week 26
Description: Maximum Total Daily Number of Self-Reported Spray Doses
Time Frame: Week 26
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 129 | 137
Number of sprays | 8.1 (7.30) | 7.9 (7.81)

96. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 1
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 1
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 512 | 502
Number of sprays | 6.0 (7.11) | 4.8 (4.93)

97. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 2
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 2
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 492 | 486
Number of sprays | 4.8 (6.13) | 3.4 (3.42)

98. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 3
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 3
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 467 | 462
Number of sprays | 4.3 (4.93) | 3.1 (2.87)

99. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 4
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 4
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 449 | 444
Number of sprays | 4.1 (4.49) | 3.0 (3.05)

100. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 5
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 5
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 423 | 428
Number of sprays | 3.7 (3.73) | 2.8 (3.25)

101. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 6
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 6
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 406 | 412
Number of sprays | 3.7 (4.23) | 2.7 (2.33)

102. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 7
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 7
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 392 | 387
Number of sprays | 3.6 (4.88) | 2.9 (4.14)

103. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 8
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 8
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 378 | 377
Number of sprays | 3.3 (3.31) | 2.6 (2.67)

104. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 9
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 9
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 356 | 362
Number of sprays | 3.3 (3.52) | 2.3 (2.13)

105. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 10
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 10
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 336 | 337
Number of sprays | 3.2 (3.28) | 2.3 (2.19)

106. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 11
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 11
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 317 | 329
Number of sprays | 3.0 (2.65) | 2.2 (2.00)

107. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 12
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 12
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 306 | 332
Number of sprays | 2.8 (2.84) | 2.0 (1.78)

108. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 13
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 13
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 240 | 251
Number of sprays | 2.7 (2.65) | 2.2 (1.72)

109. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 14
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 14
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 223 | 237
Number of sprays | 2.9 (2.69) | 2.2 (2.28)

110. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 15
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 15
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 213 | 228
Number of sprays | 2.6 (2.30) | 2.4 (3.38)

111. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 16
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 16
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 206 | 218
Number of sprays | 2.7 (3.24) | 2.1 (2.30)

112. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 17
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 17
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 189 | 194
Number of sprays | 2.5 (2.75) | 2.1 (1.72)

113. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 18
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 18
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 182 | 192
Number of sprays | 2.4 (2.22) | 2.3 (2.68)

114. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 19
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 19
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 171 | 180
Number of sprays | 2.6 (3.02) | 2.3 (2.34)

115. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 20
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 20
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 173 | 174
Number of sprays | 2.4 (2.56) | 2.0 (1.99)

116. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 21
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 21
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 164 | 161
Number of sprays | 2.3 (2.52) | 2.1 (2.10)

117. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 22
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 22
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 155 | 158
Number of sprays | 2.3 (2.86) | 2.0 (2.03)

118. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 23
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 23
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 147 | 155
Number of sprays | 2.1 (1.92) | 2.0 (2.23)

119. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 24
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 24
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 139 | 143
Number of sprays | 2.4 (4.23) | 1.9 (2.42)

120. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 25
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 25
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 142 | 143
Number of sprays | 2.0 (2.33) | 1.8 (2.09)

121. Secondary Outcome: Maximum Hourly Number of Self-Reported Spray Doses at Week 26
Description: Maximum Hourly Number of Self-Reported Spray Doses
Time Frame: Week 26
Population: Analysis was based on randomized participants who reported use data for at least 4 of the days in that week.
Measure: Mean (Standard Deviation); unit: Number of sprays
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 129 | 137
Number of sprays | 2.1 (2.59) | 1.8 (2.16)

122. Secondary Outcome: Number of Cigarettes Smoked Since Last Visit at Week 1
Description: Number of Cigarettes Smoked Since Last Visit
Time Frame: Week 1
Population: Analysis was based on randomized participants who reported non-abstinence from smoking since last visit.
Measure: Mean (Standard Deviation); unit: Number of cigarettes
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 523 | 496
Number of cigarettes | 36.2 (37.89) | 34.0 (40.57)

123. Secondary Outcome: Number of Cigarettes Smoked Since Last Visit at Week 2
Description: Number of Cigarettes Smoked Since Last Visit
Time Frame: Week 2
Population: Analysis was based on randomized participants who reported non-abstinence from smoking since last visit.
Measure: Mean (Standard Deviation); unit: Number of cigarettes
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 507 | 472
Number of cigarettes | 38.9 (44.21) | 35.8 (48.20)

124. Secondary Outcome: Number of Cigarettes Smoked Per Day at Week 4
Description: Number of Cigarettes Smoked Per Day
Time Frame: Week 4
Population: Analysis was based on randomized participants who reported non-abstinence from smoking during the preceding week.
Measure: Mean (Standard Deviation); unit: Number of cigarettes
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 451 | 430
Number of cigarettes | 7.3 (7.77) | 6.6 (8.01)

125. Secondary Outcome: Number of Cigarettes Smoked Per Day at Week 6
Description: Number of Cigarettes Smoked Per Day
Time Frame: Week 6
Population: Analysis was based on randomized participants who reported non-abstinence from smoking during the preceding week.
Measure: Mean (Standard Deviation); unit: Number of cigarettes
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 412 | 393
Number of cigarettes | 7.0 (7.63) | 6.6 (6.25)

126. Secondary Outcome: Number of Cigarettes Smoked Per Day at Week 8
Description: Number of Cigarettes Smoked Per Day
Time Frame: Week 8
Population: Analysis was based on randomized participants who reported non-abstinence from smoking during the preceding week.
Measure: Mean (Standard Deviation); unit: Number of cigarettes
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 396 | 374
Number of cigarettes | 6.8 (5.82) | 6.3 (5.93)

127. Secondary Outcome: Number of Cigarettes Smoked Per Day at Week 12
Description: Number of Cigarettes Smoked Per Day
Time Frame: Week 12
Population: Analysis was based on randomized participants who reported non-abstinence from smoking during the preceding week.
Measure: Mean (Standard Deviation); unit: Number of cigarettes
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 362 | 339
Number of cigarettes | 7.1 (5.94) | 7.5 (8.25)

128. Secondary Outcome: Number of Cigarettes Smoked Per Day at Week 16
Description: Number of Cigarettes Smoked Per Day
Time Frame: Week 16
Population: Analysis was based on randomized participants who reported non-abstinence from smoking during the preceding week.
Measure: Mean (Standard Deviation); unit: Number of cigarettes
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 316 | 315
Number of cigarettes | 7.7 (7.71) | 7.3 (6.60)

129. Secondary Outcome: Number of Cigarettes Smoked Per Day at Week 20
Description: Number of Cigarettes Smoked Per Day
Time Frame: Week 20
Population: Analysis was based on randomized participants who reported non-abstinence from smoking during the preceding week.
Measure: Mean (Standard Deviation); unit: Number of cigarettes
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 293 | 293
Number of cigarettes | 7.0 (7.50) | 7.2 (5.90)

130. Secondary Outcome: Number of Cigarettes Smoked Per Day at Week 26
Description: Number of Cigarettes Smoked Per Day
Time Frame: Week 26
Population: Analysis was based on randomized participants who reported non-abstinence from smoking during the preceding week.
Measure: Mean (Standard Deviation); unit: Number of cigarettes
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 298 | 279
Number of cigarettes | 7.2 (6.06) | 7.5 (6.71)

131. Secondary Outcome: Percentage Distribution of the Participant Score for Overall Product Rating at Week 1
Description: Participants were asked to rate the investigational product on a 10-point scale of 1 - 10 (where 1=very poor and 10=excellent).
Time Frame: Week 1
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 554 | 543
Percentage of Participants
  1 (Very Poor) | 3.2 | 1.8
  2 | 3.1 | 2.6
  3 | 2.7 | 3.9
  4 | 6.0 | 5.2
  5 | 18.6 | 16.0
  6 | 9.2 | 8.5
  7 | 18.6 | 18.8
  8 | 20.0 | 21.2
  9 | 6.7 | 7.9
  10 (Excellent) | 11.9 | 14.2

132. Secondary Outcome: Percentage Distribution of the Participant Score for Overall Product Rating at Week 6
Description: as for outcome 131
Time Frame: Week 6
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 470 | 467
Percentage of Participants
  1 (Very Poor) | 5.3 | 2.4
  2 | 2.1 | 3.0
  3 | 4.5 | 3.4
  4 | 5.1 | 3.2
  5 | 14.9 | 12.6
  6 | 8.9 | 10.3
  7 | 18.7 | 17.8
  8 | 22.3 | 21.4
  9 | 8.3 | 10.3
  10 (Excellent) | 9.8 | 15.6

133. Secondary Outcome: Percentage Distribution of the Participant Score for Overall Product Rating at Week 12
Description: as for outcome 131
Time Frame: Week 12
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 402 | 428
Percentage of Participants
  1 (Very Poor) | 5.5 | 3.5
  2 | 3.5 | 2.3
  3 | 3.7 | 3.3
  4 | 3.7 | 2.1
  5 | 11.4 | 12.4
  6 | 10.0 | 6.8
  7 | 16.7 | 14.0
  8 | 20.4 | 23.6
  9 | 10.9 | 11.0
  10 (Excellent) | 14.2 | 21.0

134. Secondary Outcome: Percentage Distribution of the Participant Score for Product Effectiveness in Dealing With Desire/Urge to Smoke at Week 1
Description: Participants were asked to rate the product in its effectiveness for dealing with desire/urge to smoke on a 5-point scale of 1 - 5 (where 1=not all effective and 5=extremely effective).
Time Frame: Week 1
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 554 | 543
Percentage of Participants
  Not at all effective (1) | 8.7 | 4.2
  Somewhat effective (2) | 27.8 | 20.8
  Moderately effective (3) | 34.5 | 32.4
  Very effective (4) | 23.3 | 29.8
  Extremely effective (5) | 5.8 | 12.7

135. Secondary Outcome: Percentage Distribution of the Participant Score for Product Effectiveness in Dealing With Desire/Urge to Smoke at Week 6
Description: as for outcome 134
Time Frame: Week 6
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 470 | 467
Percentage of Participants
  Not at all effective (1) | 11.7 | 5.4
  Somewhat effective (2) | 26.8 | 19.5
  Moderately effective (3) | 31.7 | 32.5
  Very effective (4) | 23.0 | 31.0
  Extremely effective (5) | 6.8 | 11.6

136. Secondary Outcome: Percentage Distribution of the Participant Score for Product Effectiveness in Dealing With Desire/Urge to Smoke at Week 12
Description: as for outcome 134
Time Frame: Week 12
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 402 | 428
Percentage of Participants
  Not at all effective (1) | 12.7 | 6.8
  Somewhat effective (2) | 20.1 | 17.1
  Moderately effective (3) | 32.1 | 29.7
  Very effective (4) | 25.6 | 28.7
  Extremely effective (5) | 9.5 | 17.8

137. Secondary Outcome: Percentage Distribution of the Participant Score for Speed of Action of the Product at Week 1
Description: Participants were asked to rate the speed of action of the product on a 9-point scale of 1 - 9 (where 1=extremely slow and 9=extremely fast).
Time Frame: Week 1
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 554 | 543
Percentage of Participants
  Extremely slow (1) | 4.7 | 1.8
  Very slow (2) | 2.7 | 1.5
  Moderately slow (3) | 4.0 | 2.0
  Slightly slow (4) | 6.0 | 2.8
  Neither fast nor slow (5) | 21.8 | 14.9
  Sightly fast (6) | 10.5 | 11.8
  Moderately fast (7) | 24.2 | 24.7
  Very fast (8) | 17.9 | 24.9
  Extremely fast (9) | 8.3 | 15.7

138. Secondary Outcome: Percentage Distribution of the Participant Score for Speed of Action of the Product at Week 6
Description: as for outcome 137
Time Frame: Week 6
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 470 | 467
Percentage of Participants
  Extremely slow (1) | 5.5 | 2.8
  Very slow (2) | 4.9 | 2.4
  Moderately slow (3) | 4.7 | 3.9
  Slightly slow (4) | 4.7 | 3.6
  Neither fast nor slow (5) | 20.2 | 13.3
  Sightly fast (6) | 11.9 | 9.2
  Moderately fast (7) | 24.3 | 25.3
  Very fast (8) | 18.3 | 25.1
  Extremely fast (9) | 5.5 | 14.6

139. Secondary Outcome: Percentage Distribution of the Participant Score for Speed of Action of the Product at Week 12
Description: as for outcome 137
Time Frame: Week 12
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 402 | 428
Percentage of Participants
  Extremely slow (1) | 5.5 | 4.0
  Very slow (2) | 3.5 | 1.6
  Moderately slow (3) | 4.2 | 2.6
  Slightly slow (4) | 4.7 | 3.3
  Neither fast nor slow (5) | 19.4 | 14.7
  Sightly fast (6) | 8.5 | 8.6
  Moderately fast (7) | 28.4 | 21.7
  Very fast (8) | 17.9 | 28.3
  Extremely fast (9) | 8.0 | 15.2

140. Secondary Outcome: Percentage Distribution of the Participant Score for Change of Opinion at Week 1 Concerning Product Compared to When First Used Product
Description: Participants were asked to rate their change of opinion concerning product compared to when first used product on a 5-point scale of 1 - 5 (where 1=I like it much less now and 5=I like it much more now).
Time Frame: Week 1
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 554 | 543
Percentage of Participants
  I like it much less now (1) | 2.5 | 1.7
  I like it slightly less now (2) | 4.3 | 4.8
  I like it about the same (3) | 50.9 | 44.8
  I like it slightly more now (4) | 26.4 | 28.9
  I like it much more now (5) | 15.9 | 19.9

141. Secondary Outcome: Percentage Distribution of the Participant Score for Change of Opinion at Week 6 Concerning Product Compared to When First Used Product
Description: as for outcome 140
Time Frame: Week 6
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 470 | 467
Percentage of Participants
  I like it much less now (1) | 4.7 | 4.3
  I like it slightly less now (2) | 11.9 | 7.7
  I like it about the same (3) | 47.9 | 46.9
  I like it slightly more now (4) | 22.3 | 22.9
  I like it much more now (5) | 13.2 | 18.2

142. Secondary Outcome: Percentage Distribution of the Participant Score for Change of Opinion at Week 12 Concerning Product Compared to When First Used Product
Description: as for outcome 140
Time Frame: Week 12
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 402 | 428
Percentage of Participants
  I like it much less now (1) | 9.0 | 6.5
  I like it slightly less now (2) | 9.0 | 8.4
  I like it about the same (3) | 46.0 | 44.6
  I like it slightly more now (4) | 18.7 | 20.1
  I like it much more now (5) | 17.4 | 20.3

143. Secondary Outcome: Percentage Distribution of the Participant Score for Product Convenience at Week 1
Description: Participants were asked to rate the product convenience on a 5-point scale of 1 - 5 (where 1=not at all convenient and 5=extremely convenient).
Time Frame: Week 1
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 554 | 543
Percentage of Participants
  Not at all convenient (1) | 0.9 | 0.2
  Somewhat convenient (2) | 3.2 | 3.7
  Moderately convenient (3) | 10.1 | 10.1
  Very convenient (4) | 45.1 | 41.6
  Extremely convenient (5) | 40.6 | 44.4

144. Secondary Outcome: Percentage Distribution of the Participant Score for Product Convenience at Week 6
Description: as for outcome 143
Time Frame: Week 6
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 470 | 467
Percentage of Participants
  Not at all convenient (1) | 0.9 | 0.4
  Somewhat convenient (2) | 4.7 | 3.4
  Moderately convenient (3) | 8.7 | 8.4
  Very convenient (4) | 46.2 | 50.1
  Extremely convenient (5) | 39.6 | 37.7

145. Secondary Outcome: Percentage Distribution of the Participant Score for Product Convenience at Week 12
Description: as for outcome 143
Time Frame: Week 12
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 402 | 428
Percentage of Participants
  Not at all convenient (1) | 1.5 | 0.2
  Somewhat convenient (2) | 3.0 | 4.0
  Moderately convenient (3) | 9.0 | 9.1
  Very convenient (4) | 48.0 | 44.2
  Extremely convenient (5) | 38.6 | 42.5

146. Secondary Outcome: Systolic Blood Pressure at Week 1
Description: Systolic blood pressure (mm Hg)
Time Frame: Week 1
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 562 | 554
mm Hg | 123.7 (15.54) | 124.7 (15.84)

147. Secondary Outcome: Systolic Blood Pressure at Week 2
Description: Systolic blood pressure (mm Hg)
Time Frame: Week 2
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 546 | 542
mm Hg | 123.3 (15.42) | 123.7 (15.50)

148. Secondary Outcome: Systolic Blood Pressure at Week 4
Description: Systolic blood pressure (mm Hg)
Time Frame: Week 4
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 504 | 514
mm Hg | 122.5 (15.29) | 122.9 (15.55)

149. Secondary Outcome: Systolic Blood Pressure at Week 6
Description: Systolic blood pressure (mm Hg)
Time Frame: Week 6
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 475 | 476
mm Hg | 122.3 (14.05) | 122.4 (15.04)

150. Secondary Outcome: Systolic Blood Pressure at Week 8
Description: Systolic blood pressure (mm Hg)
Time Frame: Week 8
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 459 | 457
mm Hg | 122.0 (14.52) | 122.7 (14.86)

151. Secondary Outcome: Systolic Blood Pressure at Week 12
Description: Systolic blood pressure (mm Hg)
Time Frame: Week 12
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 418 | 434
mm Hg | 121.8 (15.02) | 122.7 (15.81)

152. Secondary Outcome: Systolic Blood Pressure at Week 16
Description: Systolic blood pressure (mm Hg)
Time Frame: Week 16
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 378 | 402
mm Hg | 122.3 (14.94) | 122.8 (15.25)

153. Secondary Outcome: Systolic Blood Pressure at Week 20
Description: Systolic blood pressure (mm Hg)
Time Frame: Week 20
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 355 | 385
mm Hg | 122.4 (15.40) | 123.2 (15.41)

154. Secondary Outcome: Systolic Blood Pressure at Week 26
Description: Systolic blood pressure (mm Hg)
Time Frame: Week 26
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 354 | 365
mm Hg | 123.2 (14.44) | 124.8 (15.07)

155. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 1
Description: Change from baseline in systolic blood pressure (mm Hg)
Time Frame: Baseline to Week 1
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 562 | 554
mm Hg | -0.2 (13.49) | 0.2 (13.94)

156. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 2
Description: Change from baseline in systolic blood pressure (mm Hg)
Time Frame: Baseline to Week 2
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 546 | 542
mm Hg | -0.7 (14.06) | -0.7 (13.43)

157. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 4
Description: Change from baseline in systolic blood pressure (mm Hg)
Time Frame: Baseline to Week 4
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 504 | 514
mm Hg | -1.8 (14.59) | -1.9 (14.52)

158. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 6
Description: Change from baseline in systolic blood pressure (mm Hg)
Time Frame: Baseline to Week 6
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 475 | 476
mm Hg | -2.0 (14.80) | -2.2 (13.90)

159. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 8
Description: Change from baseline in systolic blood pressure (mm Hg)
Time Frame: Baseline to Week 8
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 459 | 457
mm Hg | -1.8 (15.26) | -2.2 (14.61)

160. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 12
Description: Change from baseline in systolic blood pressure (mm Hg)
Time Frame: Baseline to Week 12
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 418 | 434
mm Hg | -2.2 (15.75) | -2.4 (15.01)

161. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 16
Description: Change from baseline in systolic blood pressure (mm Hg)
Time Frame: Baseline to Week 16
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 378 | 402
mm Hg | -1.8 (14.95) | -2.8 (15.57)

162. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 20
Description: Change from baseline in systolic blood pressure (mm Hg)
Time Frame: Baseline to Week 20
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 355 | 385
mm Hg | -1.7 (15.15) | -2.0 (16.18)

163. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 26
Description: Change from baseline in systolic blood pressure (mm Hg)
Time Frame: Baseline to Week 26
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 354 | 365
mm Hg | -0.6 (14.61) | -0.6 (15.37)

164. Secondary Outcome: Diastolic Blood Pressure at Week 1
Description: Diastolic blood pressure (mm Hg)
Time Frame: Week 1
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 562 | 554
mm Hg | 77.3 (9.54) | 78.0 (9.99)

165. Secondary Outcome: Diastolic Blood Pressure at Week 2
Description: Diastolic blood pressure (mm Hg)
Time Frame: Week 2
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 546 | 542
mm Hg | 76.7 (9.72) | 78.0 (10.03)

166. Secondary Outcome: Diastolic Blood Pressure at Week 4
Description: Diastolic blood pressure (mm Hg)
Time Frame: Week 4
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 504 | 514
mm Hg | 76.9 (9.58) | 77.6 (9.86)

167. Secondary Outcome: Diastolic Blood Pressure at Week 6
Description: Diastolic blood pressure (mm Hg)
Time Frame: Week 6
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 475 | 476
mm Hg | 76.6 (9.86) | 76.5 (9.49)

168. Secondary Outcome: Diastolic Blood Pressure at Week 8
Description: Diastolic blood pressure (mm Hg)
Time Frame: Week 8
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 459 | 457
mm Hg | 76.5 (9.82) | 77.3 (9.35)

169. Secondary Outcome: Diastolic Blood Pressure at Week 12
Description: Diastolic blood pressure (mm Hg)
Time Frame: Week 12
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 418 | 434
mm Hg | 76.6 (10.12) | 77.4 (10.25)

170. Secondary Outcome: Diastolic Blood Pressure at Week 16
Description: Diastolic blood pressure (mm Hg)
Time Frame: Week 16
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 378 | 402
mm Hg | 76.4 (9.43) | 77.0 (10.10)

171. Secondary Outcome: Diastolic Blood Pressure at Week 20
Description: Diastolic blood pressure (mm Hg)
Time Frame: Week 20
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 355 | 385
mm Hg | 76.3 (9.91) | 76.8 (10.50)

172. Secondary Outcome: Diastolic Blood Pressure at Week 26
Description: Diastolic blood pressure (mm Hg)
Time Frame: Week 26
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 354 | 365
mm Hg | 76.9 (9.21) | 78.1 (10.13)

173. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 1
Description: Change from baseline in diastolic blood pressure (mm Hg)
Time Frame: Baseline to Week 1
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 562 | 554
mm Hg | 0.1 (8.98) | 0.5 (9.13)

174. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 2
Description: Change from baseline in diastolic blood pressure (mm Hg)
Time Frame: Baseline to Week 2
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 546 | 542
mm Hg | -0.4 (9.05) | 0.4 (9.27)

175. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 4
Description: Change from baseline in diastolic blood pressure (mm Hg)
Time Frame: Baseline to Week 4
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 504 | 514
mm Hg | -0.3 (9.58) | -0.1 (9.38)

176. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 6
Description: Change from baseline in diastolic blood pressure (mm Hg)
Time Frame: Baseline to Week 6
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 475 | 476
mm Hg | -0.6 (9.87) | -1.0 (9.37)

177. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 8
Description: Change from baseline in diastolic blood pressure (mm Hg)
Time Frame: Baseline to Week 8
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 459 | 457
mm Hg | -0.4 (10.10) | -0.1 (10.39)

178. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 12
Description: Change from baseline in diastolic blood pressure (mm Hg)
Time Frame: Baseline to Week 12
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 418 | 434
mm Hg | -0.4 (10.06) | -0.4 (10.28)

179. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 16
Description: Change from baseline in diastolic blood pressure (mm Hg)
Time Frame: Baseline to Week 16
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 378 | 402
mm Hg | -0.6 (10.19) | -0.8 (9.86)

180. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 20
Description: Change from baseline in diastolic blood pressure (mm Hg)
Time Frame: Baseline to Week 20
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 355 | 385
mm Hg | -0.8 (10.07) | -0.5 (10.69)

181. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 26
Description: Change from baseline in diastolic blood pressure (mm Hg)
Time Frame: Baseline to Week 26
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 354 | 365
mm Hg | -0.1 (10.13) | 0.7 (10.71)

182. Secondary Outcome: Pulse at Week 1
Description: Pulse (beats per minute)
Time Frame: Week 1
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 562 | 554
beats per minute | 76.1 (11.92) | 76.8 (11.45)

183. Secondary Outcome: Pulse at Week 2
Description: Pulse (beats per minute)
Time Frame: Week 2
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 546 | 542
beats per minute | 75.9 (11.82) | 76.5 (11.64)

184. Secondary Outcome: Pulse at Week 4
Description: Pulse (beats per minute)
Time Frame: Week 4
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 504 | 514
beats per minute | 75.6 (11.77) | 77.0 (11.72)

185. Secondary Outcome: Pulse at Week 6
Description: Pulse (beats per minute)
Time Frame: Week 6
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 474 | 475
beats per minute | 75.3 (11.41) | 75.2 (11.37)

186. Secondary Outcome: Pulse at Week 8
Description: Pulse (beats per minute)
Time Frame: Week 8
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 459 | 456
beats per minute | 75.4 (11.69) | 77.3 (11.27)

187. Secondary Outcome: Pulse at Week 12
Description: Pulse (beats per minute)
Time Frame: Week 12
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 417 | 434
beats per minute | 75.1 (11.46) | 76.1 (11.02)

188. Secondary Outcome: Pulse at Week 16
Description: Pulse (beats per minute)
Time Frame: Week 16
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 378 | 402
beats per minute | 76.9 (11.94) | 76.2 (11.46)

189. Secondary Outcome: Pulse at Week 20
Description: Pulse (beats per minute)
Time Frame: Week 20
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 355 | 385
beats per minute | 76.4 (11.70) | 76.2 (11.58)

190. Secondary Outcome: Pulse at Week 26
Description: Pulse (beats per minute)
Time Frame: Week 26
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 354 | 365
beats per minute | 76.9 (11.98) | 76.0 (10.85)

191. Secondary Outcome: Change From Baseline in Pulse at Week 1
Description: Change from baseline in pulse (beats per minute)
Time Frame: Baseline to Week 1
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 562 | 554
beats per minute | 1.4 (10.69) | 2.0 (10.80)

192. Secondary Outcome: Change From Baseline in Pulse at Week 2
Description: Change from baseline in pulse (beats per minute)
Time Frame: Baseline to Week 2
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 546 | 542
beats per minute | 1.2 (10.75) | 1.8 (10.95)

193. Secondary Outcome: Change From Baseline in Pulse at Week 4
Description: Change from baseline in pulse (beats per minute)
Time Frame: Baseline to Week 4
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 504 | 514
beats per minute | 1.3 (11.42) | 2.4 (11.51)

194. Secondary Outcome: Change From Baseline in Pulse at Week 6
Description: Change from baseline in pulse (beats per minute)
Time Frame: Baseline to Week 6
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 474 | 475
beats per minute | 1.0 (11.23) | 0.7 (11.44)

195. Secondary Outcome: Change From Baseline in Pulse at Week 8
Description: Change from baseline in pulse (beats per minute)
Time Frame: Baseline to Week 8
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 459 | 456
beats per minute | 1.2 (11.51) | 2.7 (11.96)

196. Secondary Outcome: Change From Baseline in Pulse at Week 12
Description: Change from baseline in pulse (beats per minute)
Time Frame: Baseline to Week 12
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 417 | 434
beats per minute | 0.9 (11.09) | 1.8 (10.84)

197. Secondary Outcome: Change From Baseline in Pulse at Week 16
Description: Change from baseline in pulse (beats per minute)
Time Frame: Baseline to Week 16
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 378 | 402
beats per minute | 2.8 (11.58) | 1.9 (11.50)

198. Secondary Outcome: Change From Baseline in Pulse at Week 20
Description: Change from baseline in pulse (beats per minute)
Time Frame: Baseline to Week 20
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 355 | 385
beats per minute | 2.7 (11.25) | 2.0 (10.96)

199. Secondary Outcome: Change From Baseline in Pulse at Week 26
Description: Change from baseline in pulse (beats per minute)
Time Frame: Baseline to Week 26
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 354 | 365
beats per minute | 3.2 (11.16) | 1.8 (11.29)

200. Secondary Outcome: Percentage of Participants With New or Worsened Conditions in Lips/Labial Mucosa at Week 6 or When Withdrawn From Study
Description: Visual mouth inspection (VMI) performed at the site or local dental office by a licensed dentist or an examiner such as a dental hygienist with documented training in oral clinical exams. Extraoral and intraoral tissues were examined. Abnormalities were recorded; it was determined if abnormalities were new or had worsened since baseline VMI findings.
Time Frame: Week 6 or when withdrawn from study
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 495 | 495
Percentage of Participants | 0.4 | 1.0

201. Secondary Outcome: Percentage of Participants With New or Worsened Conditions in Buccal Mucosa at Week 6 or When Withdrawn From Study
Description: as for outcome 200
Time Frame: Week 6 or when withdrawn from study
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 495 | 495
Percentage of Participants | 1.2 | 1.6

202. Secondary Outcome: Percentage of Participants With New or Worsened Conditions in Mucobuccal Fold at Week 6 or When Withdrawn From Study
Description: as for outcome 200
Time Frame: Week 6 or when withdrawn from study
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 495 | 494
Percentage of Participants | 0.2 | 0.0

203. Secondary Outcome: Percentage of Participants With New or Worsened Conditions in Sublingual Mucosa at Week 6 or When Withdrawn From Study
Description: as for outcome 200
Time Frame: Week 6 or when withdrawn from study
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 495 | 495
Percentage of Participants | 0.0 | 0.0

204. Secondary Outcome: Percentage of Participants With New or Worsened Conditions in Gingiva at Week 6 or When Withdrawn From Study
Description: as for outcome 200
Time Frame: Week 6 or when withdrawn from study
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 495 | 495
Percentage of Participants | 0.2 | 1.0

205. Secondary Outcome: Percentage of Participants With New or Worsened Conditions in Tongue at Week 6 or When Withdrawn From Study
Description: as for outcome 200
Time Frame: Week 6 or when withdrawn from study
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 495 | 495
Percentage of Participants | 0.8 | 0.8

206. Secondary Outcome: Percentage of Participants With New or Worsened Conditions in Hard/Soft Palate at Week 6 or When Withdrawn From Study
Description: as for outcome 200
Time Frame: Week 6 or when withdrawn from study
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 495 | 495
Percentage of Participants | 0.4 | 1.0

207. Secondary Outcome: Percentage of Participants With New or Worsened Conditions in Uvula/Oropharynx at Week 6 or When Withdrawn From Study
Description: as for outcome 200
Time Frame: Week 6 or when withdrawn from study
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 495 | 495
Percentage of Participants | 0.4 | 0.2

208. Secondary Outcome: Percentage of Participants With New or Worsened Conditions in Visual Mouth Inspection Overall at Week 6 or When Withdrawn From Study
Description: as for outcome 200
Time Frame: Week 6 or when withdrawn from study
Population: Analysis was based on the Safety Analysis Set which included all randomized participants who received study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 495 | 495
Percentage of Participants | 1.8 | 3.6

209. Secondary Outcome: Change From Baseline in Body Weight at Week 6
Description: Change from baseline in body weight
Time Frame: Baseline to Week 6
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 471 | 472
pounds | 0.5 (5.73) | 0.7 (6.29)

210. Secondary Outcome: Change From Baseline in Body Weight at Week 12
Description: Change from baseline in body weight
Time Frame: Baseline to Week 12
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 411 | 432
pounds | -0.3 (7.40) | 0.4 (6.89)

211. Secondary Outcome: Change From Baseline in Body Weight at Week 26
Description: Change from baseline in body weight
Time Frame: Baseline to Week 26
Population: Analysis was based on the Full Analysis Set which included all randomized participants.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 351 | 366
pounds | -0.2 (11.07) | 1.0 (8.43)

212. Secondary Outcome: Change From Baseline in Body Weight at Week 6 in Participants Verified Continuously Abstinent From Smoking From the Week 2 Visit
Description: Change from baseline in body weight
Time Frame: Baseline to Week 6
Population: Analysis was based on randomized participants verified continuously abstinent from smoking since the Week 2 visit.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 14 | 30
pounds | 3.6 (5.93) | 3.7 (5.79)
Statistical Analysis 1: Comparison: Placebo vs Nicotine; The null hypothesis was no difference in mean change from baseline in body weight between treatments. The alternative hypothesis was a difference in mean change from baseline in body weight between treatments; Test type: Superiority; p = 0.558, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment, baseline smoking category, study site, and baseline weight were factors; Least Squares Mean Difference = 0.99, 95% CI 2-sided [-2.42 to 4.41], Standard Error of Mean 1.679 — Least Squares Mean Difference = Nicotine - Placebo

213. Secondary Outcome: Change From Baseline in Body Weight at Week 12 in Participants Verified Continuously Abstinent From Smoking From the Week 2 Visit
Description: Change from baseline in body weight
Time Frame: Baseline to Week 12
Population: Analysis was based on randomized participants verified continuously abstinent from smoking since the Week 2 visit.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 8 | 24
pounds | 4.2 (8.89) | 6.4 (6.92)
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 212, analysis 1]; Test type: Superiority; p = 0.383, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment, baseline smoking category, study site, and baseline weight were factors; Least Squares Mean Difference = 3.04, 95% CI 2-sided [-4.03 to 10.11], Standard Error of Mean 3.409 — Least Squares Mean Difference = Nicotine - Placebo

214. Secondary Outcome: Change From Baseline in Body Weight at Week 26 in Participants Verified Continuously Abstinent From Smoking From the Week 2 Visit
Description: Change from baseline in body weight
Time Frame: Baseline to Week 26
Population: Analysis was based on randomized participants verified continuously abstinent from smoking since the Week 2 visit.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 6 | 20
pounds | 2.5 (5.67) | 9.3 (9.52)
Statistical Analysis 1: Comparison: Placebo vs Nicotine; [analysis description as in outcome 212, analysis 1]; Test type: Superiority; p = 0.138, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment, baseline smoking category, study site, and baseline weight were factors; Least Squares Mean Difference = 7.13, 95% CI 2-sided [-2.56 to 16.83], Standard Error of Mean 4.573 — Least Squares Mean Difference = Nicotine - Placebo

ADVERSE EVENTS:
Time Frame: Through 26-week end-of-study visit or through early termination visit; + up to 30 days for unresolved adverse events; +30 days for serious adverse events
Description: AEs were systematically collected during the study. AEs that were unresolved upon completion or termination from the study were followed for up to 30 calendar days until the event or its sequelae resolved or stabilized. Serious AEs were collected through 30 calendar days after the participant's last study visit.
Arm/Group | Placebo | Nicotine
Serious Adverse Events (participants affected / at risk) | 14/601 | 20/597
Other Adverse Events (participants affected / at risk) | 140/601 | 349/597
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=601) | Nicotine (N=597)
Angina Unstable (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Secondary Adrenocortical Insufficiency (Endocrine disorders) | 0 | 1
Blindness Unilateral (Eye disorders) | 0 | 1
Retinal Oedema (Eye disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Sudden Death (General disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Abdominal Abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Clostridium Difficile Infection (Infections and infestations) | 1 | 0
Device Related Infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Localised Infection (Infections and infestations) | 0 | 1
Periodontitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Post Procedural Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Postoperative Ileus (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Sternal Fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Bipolar Disorder (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Substance Abuse (Psychiatric disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 2
Renal Injury (Renal and urinary disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic Foot (Skin and subcutaneous tissue disorders) | 0 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=601) | Nicotine (N=597)
Nausea (Gastrointestinal disorders) | 26 | 59
Nasopharyngitis (Infections and infestations) | 22 | 35
Upper Respiratory Tract Infection (Infections and infestations) | 23 | 35
Headache (Nervous system disorders) | 38 | 48
Hiccups (Respiratory, thoracic and mediastinal disorders) | 47 | 252
Hypertension (Vascular disorders) | 18 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submission for publication, PI was to provide sponsor with ≥ 60 days for publication review. No publication that included sponsor confidential information was to be submitted without sponsor's consent. If requested, the PI was to withhold publication for up to 60 additional days to allow for patent application filing. First publication of study results was to be a joint, multicenter publication; if not submitted within 6 months after end of study, the PI may publish the site results.